CLINICAL TRIAL: NCT01337687
Title: Intranasal Oxytocin for the Treatment of Autism Spectrum Disorders
Acronym: INOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Eric Hollander, Clinical Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-10-303
Record Dates: First submitted 2010-12-15; First posted 2011-04-19 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism; Autism Spectrum Disorders; Oxytocin; Hollander; ASD; Asperger Syndrome; Asperger
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental)
  Interventions: Drug: Intranasal Oxytocin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin — Oxytocin administered intranasally twice a day via 1 12 unit puff to each nostril, totaling 48 IU a day.
  Arms: Oxytocin
Drug: Placebo — Saline will be administered intranasally twice a day via 1 puff per nostril, totaling 48 IU a day.
  Arms: Placebo

SUMMARY:
Autism Spectrum Disorder (ASD) is a developmental disorder characterized by abnormalities in speech and communication, impaired social functioning and repetitive behaviors and restricted interests. Oxytocin (OT) is peptide that is known for its peripheral effects on facilitating uterine contractions and milk let-down; however, studies, mainly with rodents and non-human primates, has found that OT is involved in affiliative behaviors, including sexual behavior, mother-infant and adult-adult pair-bond formation, separation distress, and other aspects of social attachment. Moreover, OT is known to play an important role in repetitive behaviors and stress reactivity. Given that repetitive behaviors and deficits in social interaction are core symptom domains of autism, and that OT is involved in the regulation of repetitive and affiliative behaviors, it is believed that OT may play a role in the etiology of autism. Moreover, preliminary data obtained by Hollander and colleagues suggests that OT may be of value in treating core autism symptoms. Specifically, synthetic oxytocin administered via intravenous infusion to adults with autism spectrum disorders (ASD) produced significant reductions in repetitive behaviors and facilitated social cognition/memory in a double-blind, placebo-controlled cross-over laboratory challenge.

Encouraged by these findings, the primary aim of this study is to investigate the safety and therapeutic efficacy of intranasal OT in treating repetitive behaviors and social functioning/cognitive deficits in adults with ASD. This research embraces a translational approach to develop a novel treatment for core ASD symptoms; given that there are currently no Food and Drug Administration (FDA) approved medication treatments for core ASD symptoms, this research addresses an important unmet need in the field. The goal of this study is to evaluate the safety and efficacy of repeated Intranasal Oxytocin Treatment (INOT)administration in adults with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* 18 to 55 years old
* Meet Diagnostic and Statistical Manual-IV (DSM-IV), Autism Diagnostic Observation Schedule(ADOS), and Autism Diagnostic Interview-Revised (ADI-R) standards for Autism Spectrum Disorder or Aspergers Syndrome
* Have a high, normal or near normal Intelligent Quotient
* Speak and Understand English fluently

Exclusion Criteria:

* Born prior to 35 weeks gestational age
* Any primary psychiatric diagnosis other than autism at the time of screening
* Medical history of neurological disease
* Medical history of known MRI/structural lesion of the brain
* Patients who are pregnant
* With a medical condition that might interfere with the conduct of the study, confound interpretation of study results or endanger their own well being
* With evidence or history of malignancy or any significant hematological, endocrine, cardiovascular, respiratory, renal, hepatic or gastrointestinal disease
* Taking psychoactive medications
* Who plan to initiate or change nonpharmacologic interventions during the study course
* Who are unable to tolerate venipuncture procedures for blood sampling

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 33.8 [21 to 45] | 32.9 [19 to 46] | 33.2 [19.9 to 46.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement on the Clinical Global Impression-Improvement (CGI-I) Scale
Description: Rating Scale that utilizes direct observation, scales and patient report to inform clinical judgment. A form of CGI that targets social functioning will be used as the primary outcome measure. Semi-structured interview.
Time Frame: 6 Weeks
Population: Participants rated as improved on the CGI-I scale
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 10 | 9
Participants | 3 | 1

2. Secondary Outcome: Change in Obsessive- Compulsive Behavior Based on Yale Brown Obsessive Compulsive Scale (YBOCS)
Description: Clinician-Rated questionnaire measuring the time spent, distress,interference, resistance, and control in relation to obsessions and compulsions based on a 5 point scale ranging from 0-5 for each category with 0 being most desirable and 5 being least. Sub-scales are added and averaged to obtain total scores.
  -scale range (total): 0 - 40 total, 0 - 7 subclinical, 8-15 mild, 16 - 23 moderate, 24 - 31 severe, 32 - 40 extreme
  Questions are rated on a 5-point scale, 0-4, increasing in severity. Obsession Rating Subscale (5 questions, ranging from 0 - 20 total) and Compulsion Rating subscale (5 questions, ranging from 0 - 20 total) are totaled and added to obtain total scores.
  -score interpretation: Higher overall scores reflect increasing symptom severity.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale
  Baseline | 12.0 (3.9) | 10.3 (2.5)
  Week 6 | 9.4 (2.9) | 8.1 (2.5)

3. Secondary Outcome: Change in Repetitive Behavior Based Repetitive Behavior Scale - Revised (RBS-R)
Description: Subscale ranges: stereotypic behavior (0 - 27);self-injurious behavior (0 - 24); compulsive behavior (0 - 18); ritualistic/Sameness Behavior (0 - 36); restricted Interests (0 - 9).
  Higher score in all subscales reflect increasing severity. Questions rate behaviors on a 4-point scale: 0 = does not occur; 1 = occurs, mild problem; 2 = occurs, moderate problem; 3 = occurs, severe problem. Subscale scores consist of sum of ratings within each question subset.
  Lower order behaviors-- stereotypy and self-injury, higher order behaviors--compulsions, rituals /sameness, restricted interests.
  Lower Order total range: 0-51, Higher Order total range: 0-63 Stereotypic behavior and Self-injurious behavior subscales were summed to create a total range for Lower Order behavior; and Compulsive behavior, ritualistic /sameness behavior, and restricted interests subscales were summed to create a total range for Higher Order behavior.
Time Frame: Baseline, week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale
  Baseline: Higher Order | 17.0 (10.6) | 20.0 (10.8)
  Week 6:Higher Order | 17.7 (16.2) | 17.8 (13.3)
  Baseline: Lower Order | 5.8 (4.6) | 4.9 (3.7)
  Week 6: Lower Order | 2.4 (2.3) | 3.7 (2.6)

4. Secondary Outcome: Change in Facial Emotion Recognition Based on Diagnostic Analysis of Nonverbal Accuracy - 2 (DANVA-2)
Description: A clinical tool measuring emotion recognition through facial expression, voice and posture.
  1. Child faces 2 (range 0 - 100, higher values reflecting higher % of errors)
  2. Adult faces 2 (range 0 - 100, higher values reflecting higher % of errors)
  3. Child paralanguage 2 (range 0 - 100, higher values reflecting higher % of errors)
  4. Adult paralanguage 2 (range 0 - 100, higher values reflecting higher % of errors) Errors are counted and organized by pre-determined affect and intensity. Subtests considered separately.
Time Frame: baseline, week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale
  DANVA -Face Baseline | 32.6 (8.8) | 39.1 (8.4)
  DANVA- FACE Week 6 | 33.5 (6.4) | 37.4 (7.4)
  DANVA- Paralanguage Baseline | 27.8 (5.7) | 34.1 (3.0)
  DANVA- Paralanguage Week 6 | 30.5 (2.7) | 35.2 (4.7)

ADVERSE EVENTS:
Arm/Group | Oxytocin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 1/10 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=10) | Placebo (N=9)
Forgetfulness (General disorders) | 1 (2) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No